CLINICAL TRIAL: NCT00318539
Title: Quetiapine Augmentation to SRIs for Patients With Obsessive Compulsive Disorder, a Double-blind, Placebo-controlled Study
Brief Title: Addition of Quetiapine in Obsessive Compulsive Disorder - Westenberg Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1441C09907
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
Quetiapine (Seroquel ®), an atypical antipsychotic registered for use in schizophrenia, which has a very low propensity of extrapyramidal and endocrine side-effects, has also been studied as an adjunct in OCD. In an open trial, ten patients with OCD who had not responded to at least three previous treatments with a SRI at maximum dose and duration were assigned to receive quetiapine in addition to a SRI for 8 weeks. Given the efficacy of quetiapine in treatment resistant patients, and given its rapid onset of action (4-6 weeks), it is postulated that the combination of a low dose atypical antipsychotic and a standard dosage of an SRI as a treatment for patients with OCD might increase the number of responders as well as the effect size.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* All patients meet the DSM IV criteria for obsessive-compulsive disorder
* Y-BOCS score > 16 if obsessions and compulsions
* Y-BOCS score > 10 if only obsessions
* Y-BOCS score > 10 if only compulsions
* Male and female, aged between 18-70 years
* Female patients of childbearing potential must have a negative pregnancy test and use a reliable method of contraception.
* Written informed consent

Exclusion Criteria:

* Presence of any of the following DSM IV conditions; major depression (with a HDRS>15, [17 item]), bipolar disorder, schizophrenia or any other psychotic condition, tic disorder, substance related disorder during the past 6 months, epilepsy, or any structural CNS disorder or stroke within the last year.
* Evidence of clinically significant and unstable cardiovascular, gastro-intestinal, pulmonary, renal, hepatic, endocrine or haematological disorders, glaucoma, myocardial infarction within the past year, or micturition abnormalities
* Patients at risk for suicide
* Multiple serious drug allergies or known allergy for the trial compounds
* Use of antipsychotics during 6 months before the screening visit
* Use of any other psychotropic drug during 6 months before the screening visit
* Cognitive and behavioural treatment 3 months prior to the screening visit
* Any known contra-indication against citalopram or quetiapine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2003-12; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The change in Yale Brown obsessive compulsive scale (Y-BOCS) from baseline to week 10 and the number of responders are the primary efficacy parameters.
Criteria for response will be a 25% or greater change from baseline on the Y-BOCS and a final CGI rating of "much improved or "very much improved".

SECONDARY OUTCOMES:
The onset of response to treatment, using the time to a sustained response as criterion
Side effect profiles, Quality of life, Cognitive functioning

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Utrecht, Netherlands